CLINICAL TRIAL: NCT04512807
Title: Low Anti-mullerian Hormone and Pregnancy Outcome in IVF
Brief Title: AMH and Pregnancy Outcome in IVF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al Baraka Fertility Hospital (Other)
Responsible Party: Principal Investigator, Dr. Kamal Rageh, doctor , medical director, Al Baraka Fertility Hospital
Other Study IDs: Dr. Atyaf Aldawodi
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: AMH

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AMH — AMH & PREGNANCY

SUMMARY:
Anti-Mu¨llerian hormone (AMH) is an established marker of ovarian reserve (La Marca et al., 2010; Nelson et al., 2009) and predicts both high and low responses in ovarian stimulation cycles (Eldar-Geva et al., 2005; Nardo et al., 2009; Nelson et al., 2007). Presently, AMH helps clinicians counsel patients prior to IVF treatment (La Marca et al., 2011), despite the fact that it fails to predict who will become pregnant (Lamazou et al., 2011; Riggs et al., 2011). It has been demonstrated that poor responders can achieve both pregnancy and live birth (Weghofer et al., 2011). There are few studies regarding extremely low AMH concentrations and live births (Fraisse et al., 2008; Tocci et al., 2009; Weghofer et al., 2011) and they present either a small number of patients or limited data describing the groups of investigated patients. Another factor affecting pregnancy rates is endometriosis, a chronic gynaecological disease characterized by the presence of functional endometrial tissue outside the uterine cavity (Koninckx et al., 1991). Many studies have reported that pregnancy rates are lower in women with endometriosis than in controls (Gupta et al., 2008; Koninckx et al., 1991 Pellicer et al., 2000). Lower AMH serum concentrations are associated with endometriosis severity (Shebl et al., 2006). The primary objective of the present study was to assess the clinical pregnancy rates in women with extremely low AMH concentrations with respect to age.

ELIGIBILITY:
Inclusion Criteria:

Women ≥22 years age AMH is 0.5 and less Body mass index- 18.5-30 kg/m 2 The normal uterine cavity on ultrasound scan At least one good quality embryo present for transfer Women willing to comply with the clinical study protocol

Exclusion Criteria:

* Women ≥ 45 years age
* AMH >0.5
* Uterine abnormalities that can compromise the IRs (e.g., endometrial polyp, fibroids, hydrosalpinx, and adenomyosis)
* Endocrine dysfunction or organ dysfunction such as liver or kidney failure.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with low or very low AMH
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-11-25 (Estimated)

PRIMARY OUTCOMES:
pregnancy test | 2 weeks
  B-HCG
clinical pregnancy rate | 4 weeks
  fetal heart activity